CLINICAL TRIAL: NCT01222000
Title: TREATMENT OF THE RECESSIVE NONBULLOUS CONGENITAL ICHTHYOSIS BY THE EPIGALLOCATECHINE CUTANEOUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Centre Hospitalier Universitaire de Nice, Centre Hospitalier Universitaire de Nice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-PP-02
Record Dates: First submitted 2010-10-12; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Lamellar Ichthyosis
MeSH Terms: conditions — Ichthyosis, Lamellar

ARMS (2):
- right controlled against moisturizing cream (Experimental)
  Interventions: Drug: apply VEREGEN ® 10 % on a randomized area and the moisturizing cream of the other side
- left controlled against moisturizing cream (Experimental)
  Interventions: Drug: apply VEREGEN ® 10 % on a randomized area and the moisturizing cream of the other side

INTERVENTIONS:
Drug: apply VEREGEN ® 10 % on a randomized area and the moisturizing cream of the other side — After inclusion, the localization of test area will be decided and the side to treat with VEREGEN 10% will be randomized. Patient will be seen every week for 4 weeks for clinical evaluation of assessment criteria by an independent assessor. According to the randomisation he will apply VEREGEN ® 10 % on a randomized area and the moisturizing cream of the other side. If there is an improvement of at least a test zone he will enter in the follow-up period for 8 weeks.
  Arms: right controlled against moisturizing cream
Drug: apply VEREGEN ® 10 % on a randomized area and the moisturizing cream of the other side — After inclusion, the localization of test area will be decided and the side to treat with VEREGEN 10% will be randomized. Patient will be seen every week for 4 weeks for clinical evaluation of assessment criteria by an independent assessor. According to the randomisation he will apply VEREGEN ® 10 % on a randomized area and the moisturizing cream of the other side. If there is an improvement of at least a test zone he will enter in the follow-up period for 8 weeks.
  Arms: left controlled against moisturizing cream

SUMMARY:
Lamellar ichthyosis (IL) is a rare autosomal recessive genodermatosis with a defect of keratinization of the skin which results in a severe generalized cutaneous xerosis with dark brown big scales, an ectropion, an eclabion, an alopecia and a palmo-plantar keratodermia. They are due to mutations of the gene TGM1 coding for the transglutaminase keratinocyte 1 (TG1) in 1/3 of the cases. Other genes were recently identified, ABCA12 coding for the triphosphate-binding adenosine cassette A12 and FLJ39501 which codes for a protein of the cytochrome p450 ( CYP4F2).

No etiological treatment is available. Symptomatic treatment consists on twice application of emollients and keratolytic ointments which decrease the dryness of the skin and reduce scales. Oral isotretinoin is usually partially effective but is only suspensive and has numerous side effects.

Recent studies showed that the epigallocatechin-3-gallate (POLYPHENON E®), extracted from green tea increases the differentiation of the normal human keratinocytes, as showedb by the increase of the involucrine, TG1 and caspase-14 genes expression.

The main objective of this pilot study is to estimate the action and the tolerance of a daily application of topical Polyphénon E 10% ® to improve the desquamation and the cutaneous roughness of patients with lamellar ichthyosis, after 4 weeks of treatment.

The secondary objectives

* To estimate the duration of remission obtained after the treatment
* To estimate the action of cutaneous Veregen® to improve the palmar and plantar involvement.
* To estimate the action of cutaneous Veregen on the pruritus
* And to estimate the global level of acceptability by the patient of the Veregen 10 %

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes of at least 8 years and less than 65 years.
* Patients with a clinical diagnosis of LI
* Patients having at once a score of roughness and a desquamation of intensity moderated in severe (at least 2) on every side of the body,
* Patients and\or relatives / representatives of the parental authority in measure to understandand to follow the procedures of the study
* Consent of patient and\or parents / representatives of the parental authority
* Patient member to the Social Security

Exclusion Criteria:

* Patient of less than 8 years
* Pregnant, breast-feeding women or old enough to procreate without reliable medical contraception,
* Women with a positive pregnancy test,
* Transaminases > twice the normal.
* Patients with congenital ichthyosis others than LI,
* Patients with a erythrodermic composent,
* Patients affected by LI of the light gravity (score < 2 for the desquamation or the roughness) on at least a side of the body,
* Patients with secondary infection ,
* Patients with known allergy of to one of the ingredients contained in the tested product,
* Patients with specific topical treatment (for example analogues of vitamin A, vitamin D similar),
* Patients with topical keratolytic treatment (for example the urea, the hydroxy-acids) in 7 days before the beginning of the clinical trial
* Patients and\or relatives / representatives of the parental authority unable to understand and\or to follow the procedures of the study,
* Tea intake during the trail

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
action and the tolerance of a daily application of topical Polyphénon E 10% ® | 4 weeks
  The main objective of this pilot study is to estimate the action and the tolerance of a daily application of topical Polyphénon E 10% ® to improve the desquamation and the cutaneous roughness of patients with lamellar ichthyosis, after 4 weeks of treatment.

SECONDARY OUTCOMES:
severity of the palmar and plantar involvement | J28
level of pruritus | until J28
global tolerance and acceptability by the patient of the Polyphénon E ® ointment | J28
Relapse | J84

CONTACTS AND LOCATIONS:
Overall Officials: Chiaverini Christine, Dr, Principal Investigator — CHU de Nice - Service de dermatologie
Locations (1):
- Toulouse University Hospital, Dermatology Department, Toulouse, France